CLINICAL TRIAL: NCT01848600
Title: Impact of a Limitation Section on the Meta-analysis Results' Interpretation: a Randomized Controlled Trial
Brief Title: Impact of a Limitation Section on the Meta-analysis Results' Interpretation
Acronym: ILMARI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: RAV003
Record Dates: First submitted 2013-02-25; First posted 2013-05-07 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2013-01

CONDITIONS: Systematic Review With Metaanalysis
Keywords: limitation; quality; bias; meta-analysis; interpretation; abstract

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- abstract without limitation section (Experimental): the experimental arm is abstract without the limitation section
  Interventions: Behavioral: interpretation of the abstract
- abstract with limitation section (Other): the control arm is abstract with the original limitation section
  Interventions: Behavioral: interpretation of the abstract

INTERVENTIONS:
Behavioral: interpretation of the abstract — the intervention consist to interpret the results of the meta-analysis after reading the abstract.

SUMMARY:
Objective: The investigators aim to evaluate the impact of a " limitations " section in systematic review's abstract on results' interpretation by readers.

Design: Randomized ratio 1:1 controlled trial with two parallel arms. Participants will be invited to participate in an online survey.

Participants: Eligible participants are corresponding authors of randomized controlled trial published between 2010 and 2012 and referenced in pubmed Intervention: The investigators will evaluate the impact of the presence of a " limitations " section in abstract of systematic review with meta-analysis. The investigators selected abstracts of meta-analysis published in the journal Annals of Internal Medicine between 2006 and 2011.

Selected abstract will be standardised and the treatment's name hidden. The two groups of abstract will be presented as follow: 1) abstract with " limitations " section and 2) abstract without " limitations " section: the " limitations " section of the original abstract will be deleted.

Selected participants are invited by e-mail to answer the survey. After reading one abstract from his group a randomization they are invited two answer 5 questions about their interpretation of the meta-analysis's results.

DETAILED DESCRIPTION:
OBJECTIVE The aim of the study is to evaluate the impact of a " limitations " section in systematic review's abstract on results' interpretation by readers.

STUDY DESIGN The study is a randomized controlled trial with two parallel arms. The study follows the CONSORT 2010 statements Participant will be invited to participate in an on-line survey with a secured web site. Participants, after a characteristic description will be randomized in one of the two arms: 1) abstract with a " limitations " section 2) abstract without a " limitations " section.

ELIGIBILITY Eligible participants are corresponding authors of randomized trials published between 2010 and 2012 and referenced in pubmed core set journal

INTERVENTION We will evaluate the impact of the presence of a " limitations " section in abstract of systematic review with meta-analysis.

SELECTION OF ABSTRACTS We will retrieve all systematic review with meta-analysis published in the journals Annals of Internal Medicine between the years 2006 and 2012, about health care intervention with a conclusion in favor the experimental treatment or intervention. We exclude updates, diagnostical, genetical, epidemiological or economical evaluation and multiple or indirect comparisons.

MODIFICATION OF ABSTRACTS All selected abstracts will be standardised. Treatment name will be replaced with "experimental treatment A", control treatment will be replaced by "control treatment B" if necessary in the title and in the abstract.

The two groups of abstract will be presented as follow:

1. Abstract with " limitations " section
2. Abstract without " limitations " section: the " limitations " section of the original abstract will be deleted.

OUTCOMES PRIMARY OUTCOME The primary outcome will be, the readers' recommendation of the experimental treatment A

SECONDARY OUTCOMES Secondary outcomes will evaluate the interpretation of the results of the meta-analysis. The readers will answers the following questions, with the choice of answers based on a 10-point Likert scale

1. How would you rate the quality of the systematic review?
2. How confident are you in the results of this systematic review?
3. Do you consider that the experimental treatment A is a proven effective treatment?
4. How confident are you in the validity of the conclusion that the authors draw? NUMBER OF PARTICIPANT A power analysis was conducted to estimate the number of subject (participants) needed to achieve a power of 0.9 and an alpha value of 0.05 to discern a different of effect size of 0.4 between the two versions of abstract. This resulted in an estimate to the need of recruit a minimum of 133 participants in each arm, either a total of 266 participants STATISTICAL ANALYSIS We will analyze data with R project software, in intention to treat. Data for quantitative variables are expressed with medians and interquartile (IQR) ranges. Qualitative variables are expressed with frequencies and percentages and missing data Primary analysis will compare means of the primary outcome between the 2 groups with a Student t test.

ELIGIBILITY:
Inclusion Criteria:

* abstract of meta-analysis published in the journal "Annals of Internal Medicine" between 2006 and 2012, about health care intervention with a conclusion in favour the experimental treatment

Exclusion Criteria:

* updates of previously published systematic reviews,
* systematic review if diagnostic test accuracy, prognosis, epidemiologic, economics evaluation
* indirect comparison meta-analysis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-04; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
confidence in the results | 1 month
  we ask participants: "how confident are you in the results of this systematic review?"

SECONDARY OUTCOMES:
interpretation of the quality of the systematic review | 1 month
  We ask participants:
  " how would you rate the quality of the systematic review?" "how confident are you in the validity of the conclusion of the systematic review?" "how confident are you that intervention A is more beneficial than comparative intervention?" "how confident are you that the results of this systematic review could be apply in clinical practice?"

CONTACTS AND LOCATIONS:
Overall Officials: Amélie YAVCHITZ, MD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France